CLINICAL TRIAL: NCT00469157
Title: Refractive Surgery and Optive Compatibility Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovative Medical (Industry)
Responsible Party: Loren Rude, OD, TLC
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 5303
Record Dates: First submitted 2007-05-02; First posted 2007-05-04 (Estimated); Last update posted 2008-04-17 (Estimated); Status verified 2008-04

CONDITIONS: Dry Eye Syndromes
Keywords: compatibility of Optive after PRK or LASIK
MeSH Terms: conditions — Dry Eye Syndromes

ARMS (1):
- 1. (Other)
  Interventions: Drug: Optive

INTERVENTIONS:
Drug: Optive — Optive 30ml- (in the eye) Instill one in each eye twice daily starting one week after surgery

SUMMARY:
To assess the compatibility of Optive with refractive surgery (PRK and LASIK) post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 and over
* Patients undergoing refractive surgery

Exclusion Criteria:

* Concurrent ocular conditions or pathology that could affect patient's ability to complete study
* Concurrent use of topical medications other than study medications
* Use of systemic medications with ocular drying sequelae:

  * Antihistamines
  * Decongestants
  * Antispasmotics
  * Antidepressants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2007-05; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Assess compatibility | 8 months

SECONDARY OUTCOMES:
comfort | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Loren Rude, OD, Principal Investigator — TLC
Locations (1):
- TLC, Fullerton, California, United States